CLINICAL TRIAL: NCT01386632
Title: Phase II Study of DCA (Dichloroacetate) in Combination With Cisplatin and Definitive Radiation in Stage III-IV Squamous Cell Carcinoma of the Head and Neck
Brief Title: Study of DCA (Dichloroacetate) in Combination With Cisplatin and Definitive Radiation in Head and Neck Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanford Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DCA 2010
Record Dates: First submitted 2011-05-23; First posted 2011-07-01 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
Keywords: Stage III-IV Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Dichloroacetic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DCA (dichloroacetate) Treatment (Active Comparator): DCA orally 12.5mg/kg or per G-tube BID daily for 8 weeks in conjunction with Cisplatin 100 mg/m^2 IV over 30-60 minutes every 3wks X 3(Days 1, 22, and 43 of RT)and RT 70 Gy/35 -200 cGy/d x 7 weeks (35 Fractions)
  Interventions: Drug: DCA (dichloroacetate)
- Placebo (Placebo Comparator): Placebo orally or per G-tube BID for 8 weeks in conjunction with Cisplatin 100 mg/m^2 IV over 30-60 minutes every 3wks X 3(Days 1, 22, and 43 of RT)and RT 70 Gy/35 -200 cGy/d x 7 weeks (35 Fractions)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DCA (dichloroacetate) — DCA orally 12.5mg/kg PO or per G-tube BID daily for 8 weeks in conjunction with Cisplatin 100 mg/m^2 IV over 30-60minutes every 3wks X 3(Days 1, 22, and 43 of RT)and RT 70 Gy/35 -200 cGy/d x 7 weeks (35 Fractions)
  Other Names: dichloroacetate
  Arms: DCA (dichloroacetate) Treatment
Drug: Placebo — Placebo PO or per G-tube twice a day for 8 weeks given in combination with Cisplatin.
  Arms: Placebo

SUMMARY:
This will be a randomized masked placebo-controlled single-center study to evaluate the effects of Dichloroacetate (DCA) versus placebo given in combination with Cisplatin and radiation treatment in patients with Stage III-IV Squamous Cell Carcinoma of the Head and Neck (SCCHN). Fifty subjects will be enrolled and randomly assigned on a 1:1 ratio to DCA or matching placebo given with standard of care treatment consisting of Cisplatin and radiation treatment.

Patients will receive DCA/placebo PO or per G-tube twice a day for 8 weeks. The first 6 patients of the total study population will represent a safety lead-in cohort. The results of the safety lead-in of DCA/placebo in combination with Cisplatin and radiation therapy will be evaluated after the 6th patient has completed 8 weeks of therapy. Recruitment of patients will be withheld during safety data analysis.

DETAILED DESCRIPTION:
Doses for Cisplatin will be based on actual body weight taken on each day of Cisplatin therapy. DCA doses will be calculated at baseline according to actual body weight and will not change during the 8 weeks of therapy.

A careful description of the extent of the primary lesion and nodal spread will be recorded.

Dental Evaluation: Prior to treatment, patients will be evaluated by the dental service and a prophylactic cleaning/fluoride regimen instituted. A delay of at least 14 days from major surgery, including dental extractions, will be required prior to Day 1 treatment.

Airway Patency: Significant laryngeal edema has been described after the use of cisplatin containing regimens. Patients with laryngeal tumors should be considered for a prophylactic tracheostomy prior to the initiation of chemotherapy, if any possibility of airway compromise exists. Patients with laryngeal tumors experiencing respiratory stridor or compromise shortly after chemotherapy/radiotherapy administration should be rapidly evaluated for tracheostomy.

Alimentation: Significant stomatitis, mucositis and dysphagia are expected with these treatment regimens. Hospitalization may be required for symptomatic management. Pronounced weight loss is common, and adequate alimentation needs to be maintained. Early, if not pre-emptive, enteral tube feedings should be considered if difficulty is anticipated.

Compliance: The complexity of these treatment regimes and their attendant toxicity are such that compliance is of major concern. Patients expected to pose compliance problems should not be entered on this study. Patients will need to be seen at least weekly during therapy so that the toxicities can be monitored and treated.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically, cytologically confirmed and previously untreated stage 3 or 4 HNSC that recommended treatment would be concurrent cisplatin and radiation.
* Age ≥ 18 years
* ECOG performance status ≤ 2 or Karnofsky ≥70%
* Life expectancy of greater than 12 weeks.
* Patients must have normal organ and marrow function as defined below:

  * Absolute neutrophil count ≥1,500/mcL
  * Hemoglobin ≥90 g/L
  * Platelets ≥100,000/mcL
  * Total bilirubin ≤1.5 X upper limit of normal (ULN)
  * AST(SGOT) and ALT(SGPT) ≤2.5 X ULN or ≤ 5 X ULN in the presence of liver metastases
  * Creatinine ≤1.5 X institutional upper limit of normal
* The effects of DCA on the developing human fetus are unknown. For this reason and because DCA can be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (e.g.: hormonal or barrier method of birth control, abstinence)prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand the purpose of the study and the willingness to sign a written informed consent document.
* Repeat biopsy is not mandatory, but is strongly suggested. Should be performed between Day 8 and Day 15 treatments.

Exclusion Criteria:

* Patients may not be receiving any other investigational agents, chemotherapy, immunotherapy, radiotherapy, or molecular targeted agents.
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that could confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to DCA.(Cetuximab)
* Due to the possibility of peripheral sensorimotor neuropathy from DCA, the presence of grade 2 or higher peripheral neuropathy due to a prior medical condition (such as multiple sclerosis), medications, or other etiologies.
* Any psychological, familial, sociological, or geographical conditions that do not permit medical follow-up and compliance with the study protocol.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, diabetes mellitus, or psychiatric illness/social situations that would limit compliance with study requirements. Specifically, for patients who are taking either or both oral hypoglycemics and insulin for diabetes mellitus will not be eligible as DCA in combination with these agents may increase the risk of clinically significant hypoglycemia, compromising patient safety.
* Pregnant or breast-feeding women are excluded from this study because DCA is an agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with DCA, breastfeeding should be discontinued if the mother is treated with DCA.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with DCA. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy.
* Five years must have elapsed since the initial curative procedure for other malignancies, except for in situ cervical cancer, basal cell carcinoma of the skin, and localized prostate cancer after curative therapy such as surgery, or radiation.
* History of malabsorption syndrome or substantial amount of small bowels or stomach removed that may impair absorption of DCA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-05; Primary Completion 2014-08 (Actual); Study Completion 2020-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven F Powell, MD, Study Chair — Sanford Health
Locations (2):
- United States (2):
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Sanford Hematology and Oncology, Sioux Falls, South Dakota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Powell SF, Mazurczak M, Dib EG, Bleeker JS, Geeraerts LH, Tinguely M, Lohr MM, McGraw SC, Jensen AW, Ellison CA, Black LJ, Puumala SE, Reed VJ, Miskimins WK, Lee JH, Spanos WC. Phase II study of dichloroacetate, an inhibitor of pyruvate dehydrogenase, in combination with chemoradiotherapy for unresected, locally advanced head and neck squamous cell carcinoma. Invest New Drugs. 2022 Jun;40(3):622-633. doi: 10.1007/s10637-022-01235-5. Epub 2022 Mar 21. PMID 35312941

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DCA (Dichloroacetate) Treatment | Placebo
Started | 25 | 25
Completed | 20 | 21
Not Completed | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DCA (Dichloroacetate) Treatment | Placebo | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.89 (9.06) | 58.35 (8.33) | 59.62 (8.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 6 | 7
  Male | 24 | 19 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 24 | 24 | 48
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 25 | 24 | 49
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced Adverse Events During Treatment.
Description: Percentage of Participants Who Experienced Adverse Events During Treatment including but are not limited to mucositis, leucopenia, neuropathy, and treatment breaks. This will be done according to the Common Terminology Criteria for Adverse Events (CTCAE), version 4.0
Time Frame: Adverse events (AE) will be assessed from the time the subject begins the study until the 30-days after receiving the last dose of the study medication.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | DCA (Dichloroacetate) Treatment | Placebo
Number analyzed (Participants) | 25 | 25
percentage of patients | 96 [79.7 to 99.9] | 96 [79.7 to 99.9]

2. Secondary Outcome: Two-year Progression-free Survival Rate in Locally Advanced Head and Neck Squamous Cell Carcinoma in Patients Receiving Concurrent Cisplatin, Radiation Therapy, and DCA.
Description: Outcome of tumor change will be compared in two separate ways. First, change in measured tumor size at 8 weeks and 3 months will be compared using standard linear models methods (using appropriate transformation to reduce statistical skew).
  Progression was determined using RECIST 1.1 definition of 20% increase in the sum of the diameters of target lesions, in either primary or nodal lesions or the appearance of one or more new lesion(s) and/or unequivocal progression of existing non-target lesions.
Time Frame: Year 2
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | DCA (Dichloroacetate) Treatment | Placebo
Number analyzed (Participants) | 25 | 25
percentage of patients | 86.5 [72.3 to 100] | 87.5 [74.3 to 100]

3. Secondary Outcome: Two-year and Five-year Progression-free Survival Rate in Locally Advanced Head and Neck Squamous Cell Carcinoma in Patients Receiving Concurrent Cisplatin, Radiation Therapy, and DCA.
Description: Progression will be determined using RECIST 1.1 definition of 20% increase in the sum of the diameters of target lesions, in either primary or nodal lesions or the appearance of one or more new lesion(s) and/or unequivocal progression of existing non-target lesions.
Time Frame: Year 5
Reporting Status: Not Posted

4. Secondary Outcome: Local Response Rate for Locally Advanced Head and Neck Squamous Cell Carcinoma Patients Receiving Concurrent Cisplatin, Radiation Therapy, and DCA.
Time Frame: 3 months
Reporting Status: Not Posted

5. Secondary Outcome: Local Response Rate for Locally Advanced Head and Neck Squamous Cell Carcinoma Patients Receiving Concurrent Cisplatin, Radiation Therapy, and DCA.
Time Frame: 1 year
Reporting Status: Not Posted

6. Secondary Outcome: Overall Survival for Locally Advanced Head and Neck Squamous Cell Carcinoma Patients Receiving Concurrent Cisplatin, Radiation Therapy, and DCA.
Time Frame: 1 year
Reporting Status: Not Posted

7. Secondary Outcome: Overall Survival for Locally Advanced Head and Neck Squamous Cell Carcinoma Patients Receiving Concurrent Cisplatin, Radiation Therapy, and DCA.
Time Frame: 2 years
Reporting Status: Not Posted

8. Secondary Outcome: Overall Survival for Locally Advanced Head and Neck Squamous Cell Carcinoma Patients Receiving Concurrent Cisplatin, Radiation Therapy, and DCA.
Time Frame: 5 year
Reporting Status: Not Posted

9. Secondary Outcome: Health-related Quality of Life Among Study Patients by Treatment Arm.
Time Frame: Completion of Treatment
Reporting Status: Not Posted

10. Secondary Outcome: Health-related Quality of Life Among Study Patients by Treatment Arm .
Time Frame: 1 year
Reporting Status: Not Posted

11. Secondary Outcome: Health-related Quality of Life Among Study Patients by Treatment Arm.
Time Frame: 2 year
Reporting Status: Not Posted

12. Secondary Outcome: Health-related Quality of Life Among Study Patients by Treatment Arm .
Time Frame: 5 year
Reporting Status: Not Posted

13. Secondary Outcome: Immune Response and Correlate These Findings With Toxicity and Outcome (Exploratory Analysis).
Time Frame: 3 months
Reporting Status: Not Posted

14. Secondary Outcome: HPV Status- Correlate These Findings With Toxicity and Outcome (Exploratory Analysis).
Time Frame: 3 months
Reporting Status: Not Posted

15. Secondary Outcome: Relative Toxicities for Locally Advanced Head and Neck Squamous Cell Carcinoma Patients Receiving Concurrent Cisplatin, Radiation Therapy, and DCA.
Time Frame: 2 years
Reporting Status: Not Posted

16. Secondary Outcome: Relative Toxicities for Locally Advanced Head and Neck Squamous Cell Carcinoma Patients Receiving Concurrent Cisplatin, Radiation Therapy, and DCA.
Time Frame: 3 months
Reporting Status: Not Posted

17. Secondary Outcome: Relative Toxicities During Treatment for Locally Advanced Head and Neck Squamous Cell Carcinoma Patients Receiving Concurrent Cisplatin, Radiation Therapy, and DCA.
Time Frame: End of treatment
Reporting Status: Not Posted

18. Secondary Outcome: Relative Toxicities for Locally Advanced Head and Neck Squamous Cell Carcinoma Patients Receiving Concurrent Cisplatin, Radiation Therapy, and DCA.
Time Frame: 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data collected from first day of treatment to 30 days post last day of treatment, up to 2 years post treatment.
Arm/Group | DCA (Dichloroacetate) Treatment | Placebo
Serious Adverse Events (participants affected / at risk) | 8/25 | 6/25
Other Adverse Events (participants affected / at risk) | 25/25 | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DCA (Dichloroacetate) Treatment (N=25) | Placebo (N=25)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
creatinine increased (Investigations) | 0 (0) | 1 (1)
Infection and infestation-Other (Infections and infestations) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (2) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0)
Mucositis Oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DCA (Dichloroacetate) Treatment (N=25) | Placebo (N=25)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 3 (3)
Agitation (Psychiatric disorders) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 5 (5) | 5 (5)
Alkaline Phosphatase Increased (Investigations) | 2 (2) | 4 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 7 (7) | 15 (15)
Anemia (Blood and lymphatic system disorders) | 23 (23) | 23 (23)
Anorexia (Metabolism and nutrition disorders) | 23 (23) | 22 (22)
Anxiety (Psychiatric disorders) | 9 (9) | 14 (14)
Arthraligia (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 5 (5) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Blurred vision (Eye disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 19 (19) | 19 (19)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Creatinine increased (Investigations) | 7 (7) | 5 (5)
Dehydration (Metabolism and nutrition disorders) | 5 (5) | 5 (5)
Dermatitis Radiation (Injury, poisoning and procedural complications) | 17 (17) | 18 (18)
Diarrhea (Gastrointestinal disorders) | 6 (6) | 6 (6)
Dizziness (Nervous system disorders) | 8 (8) | 5 (5)
Dry Mouth (Gastrointestinal disorders) | 22 (22) | 24 (24)
Dysgeusia (Nervous system disorders) | 23 (23) | 24 (24)
Dyspepsia (Gastrointestinal disorders) | 9 (9) | 12 (12)
Dysphagia (Gastrointestinal disorders) | 20 (20) | 22 (22)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 7 (7)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 4 (4)
Edema Limbs (General disorders) | 2 (2) | 1 (1)
Fatigue (General disorders) | 22 (22) | 23 (23)
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Fever (General disorders) | 11 (11) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 8 (8) | 10 (10)
Headache (Nervous system disorders) | 0 (0) | 8 (8)
Hearing Impaired (Ear and labyrinth disorders) | 5 (5) | 3 (3)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4)
Hot Flashes (Vascular disorders) | 2 (2) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hypertension (Vascular disorders) | 10 (10) | 9 (9)
Hypoalbuminenia (Metabolism and nutrition disorders) | 12 (12) | 11 (11)
Hypocalcemia (Metabolism and nutrition disorders) | 9 (9) | 8 (8)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 8 (8) | 8 (8)
Hypomagnesemia (Metabolism and nutrition disorders) | 10 (10) | 9 (9)
Hyponatremia (Metabolism and nutrition disorders) | 20 (20) | 20 (20)
Hypotension (Vascular disorders) | 7 (7) | 1 (1)
Insomnia (Psychiatric disorders) | 18 (18) | 17 (17)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Lymphocyte count decreased (Investigations) | 19 (19) | 17 (17)
Lymphocyte count increased (Investigations) | 2 (2) | 0 (0)
Mucosal infection (Infections and infestations) | 2 (2) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 22 (22) | 23 (23)
Nausea (Gastrointestinal disorders) | 20 (20) | 20 (20)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Neutrophil count decreased (Investigations) | 18 (18) | 15 (15)
Oral pain (Gastrointestinal disorders) | 7 (7) | 6 (6)
pain (General disorders) | 4 (4) | 3 (3)
Paresthesia (Nervous system disorders) | 2 (2) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 14 (14) | 11 (11)
Platelet count decreased (Investigations) | 19 (19) | 9 (9)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 16 (16)
Tinnitus (Ear and labyrinth disorders) | 15 (15) | 21 (21)
Tremor (Nervous system disorders) | 6 (6) | 3 (3)
Vomiting (Gastrointestinal disorders) | 16 (16) | 18 (18)
Weight Loss (Investigations) | 21 (21) | 21 (21)
White blood cells decreased (Investigations) | 22 (22) | 19 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes